CLINICAL TRIAL: NCT02587546
Title: Thulium Contact Laser in the Treatment of Tumorous and Non-tumorous Laryngotracheal Stenosis
Brief Title: Thulium Contact Laser of Laryngotracheal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-thulium
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Laryngeal Carcinoma; Bilateral Vocal Cord Paresis; Subglottic Stenosis
Keywords: laryngeal carcinoma; bilateral vocal cord paralysis; laryngotracheal stenosis; laser treatment; decannulation; voice; swallowing
MeSH Terms: conditions — Laryngeal Neoplasms; Vocal Cord Paralysis | interventions — GGNBP2 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- laryngeal carcinoma (Experimental): patients with T1-T2 (some T3) laryngeal carcinoma will undergo treatment using thulium contact laser surgery - tumour resection
  Interventions: Procedure: laryngeal carcinoma
- bilateral vocal cord paralysis (Experimental): patients with bilateral vocal cord paralysis treated with partial arytenoidectomy will be treated using thulium laser surgery and laterofixation
  Interventions: Procedure: bilateral vocal cord paralysis
- subglottic stenosis (Experimental): patients with subglottic stenosis treated endoscopically (incisions and dilatation) will be treated with thulium laser surgery
  Interventions: Procedure: subglottic stenosis

INTERVENTIONS:
Procedure: laryngeal carcinoma — treatment of laryngeal carcinoma using thulium contact laser
  Arms: laryngeal carcinoma
Procedure: bilateral vocal cord paralysis — treatment of bilateral vocal cord paralysis using thulium contact laser
  Arms: bilateral vocal cord paralysis
Procedure: subglottic stenosis — treatment of subglottic stenosis using thulium contact laser
  Arms: subglottic stenosis

SUMMARY:
The purpose of the study is to compare results of the treatment of tumorous and non-tumorous laryngotracheal stenosis using thulium contact laser versus carbon dioxide laser used in the past.

DETAILED DESCRIPTION:
Laryngotracheal stenosis is a serious disease significantly worsening the quality of life. Impaired breathing often leads to tracheotomy, deterioration of the voice leads to communication problems with others and swallowing problems are often present, as well The main causes of laryngotracheal stenosis are post intubation and post tracheostomy conditions, inflammatory process (often autoimmune), tumors (mainly squamous cell carcinoma and chondroma) and trauma. Within the last years there is substantial shift in the treatment strategy from open surgery to endoscopic techniques. However, surgical treatment is often difficult due to demanding exposure of tumor and problematic margins control.

In recent years there has been a development of particular techniques of endoscopic resection of tumors and non-malignant laryngeal glottic and subglottic stenosis using a carbon dioxide (CO2) laser with promising improvement of treatment results.

However, CO2 laser has some limitations, particularly in the treatment of tumors spreading into anterior commissure, because CO2 laser beam cannot get "around the corner". Moreover, subglottic area is also difficult to be reached by CO2 laser beam. Therefore, contact laser with adjustable manipulators with possibility to bend tip of manipulator according to the actual need seems to be of some advantage.

ELIGIBILITY:
Inclusion Criteria:

1. patients with T1-T2 (some T3) laryngeal carcinoma
2. patients with bilateral vocal cord paralysis treated with partial arytenoidectomy and laterofixation
3. patients with subglottic stenosis treated endoscopically

Exclusion Criteria:

* non signing of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Percentage of carcinoma recurrence in the patient population | 36 months
  The percentage of carcinoma recurrence will be monitored and evaluated within the study subjects.

SECONDARY OUTCOMES:
Percentage of decannulation in the patient population | 36 months
  The percentage of decannulation will be monitored among the study subjects.
Voice quality (Voice Handicap Index) | 36 months
  Voice quality will be assessed according to the Voice Handicap Index, which is an acknowledged measurement tool providing precise evaluation of the condition.
Swallowing (SWAL-QOL) questionnaire | 36 months
  Swallowing will be assessed in the study group using the SWAL-QOL measurement tool (questionnaire) providing precise evaluation of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Karol Zelenik, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Warner L, Chudasama J, Kelly CG, Loughran S, McKenzie K, Wight R, Dey P. Radiotherapy versus open surgery versus endolaryngeal surgery (with or without laser) for early laryngeal squamous cell cancer. Cochrane Database Syst Rev. 2014 Dec 12;2014(12):CD002027. doi: 10.1002/14651858.CD002027.pub2. PMID 25503538
- [Background] Greulich MT, Parker NP, Lee P, Merati AL, Misono S. Voice outcomes following radiation versus laser microsurgery for T1 glottic carcinoma: systematic review and meta-analysis. Otolaryngol Head Neck Surg. 2015 May;152(5):811-9. doi: 10.1177/0194599815577103. Epub 2015 Apr 2. PMID 25837666
- [Background] Mendelsohn AH, Kiagiadaki D, Lawson G, Remacle M. CO2 laser cordectomy for glottic squamous cell carcinoma involving the anterior commissure: voice and oncologic outcomes. Eur Arch Otorhinolaryngol. 2015 Feb;272(2):413-8. doi: 10.1007/s00405-014-3368-9. Epub 2014 Oct 29. PMID 25351502
- [Background] Szakacs L, Sztano B, Matievics V, Bere Z, Bach A, Castellanos PF, Rovo L. A comparison between transoral glottis-widening techniques for bilateral vocal fold immobility. Laryngoscope. 2015 Nov;125(11):2522-9. doi: 10.1002/lary.25401. Epub 2015 Jun 8. PMID 26059854
- [Background] Riffat F, Palme CE, Veivers D. Endoscopic treatment of glottic stenosis: a report on the safety and efficacy of CO2 laser. J Laryngol Otol. 2012 May;126(5):503-5. doi: 10.1017/S002221511100301X. Epub 2011 Nov 1. PMID 22040808
- [Background] Gallo A, Pagliuca G, Greco A, Martellucci S, Mascelli A, Fusconi M, De Vincentiis M. Laryngotracheal stenosis treated with multiple surgeries: experience, results and prognostic factors in 70 patients. Acta Otorhinolaryngol Ital. 2012 Jun;32(3):182-8. PMID 22767984